CLINICAL TRIAL: NCT06564883
Title: Clinical Evaluation of Hydration and Acceptability of the Genital and Cutaneous Mucosa of a Vaginal Moisturizer in Vaginal Dryness in Menopausal Women
Brief Title: Hydration and Acceptability of the Genital and Skin Mucosa of a Vaginal Moisturizer in Menopausal Women
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BS-GIMM24
Record Dates: First submitted 2024-08-15; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Vaginismus; Vaginal Atrophy; Menopause
MeSH Terms: conditions — Vaginismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Hyaluronic Acid will applied under recommended conditions during the period of T22 ±2 days.
  Interventions: Device: 0.20% sodium hyaluronate gel

INTERVENTIONS:
Device: 0.20% sodium hyaluronate gel — Hyaluronic Acid is indicated for the relief of vaginal dryness, itching, and irritation, or the reduction of vaginal lubrication with prolonged hydration effects for up to 72 hours.
  Other Names: Hyaluronic Acid

SUMMARY:
Hyaluronic Acid is indicated for the relief of vaginal dryness, itching, and irritation, or the reduction of vaginal lubrication with prolonged hydration effects for up to 72 hours. Hyaluronic Acid promotes vaginal moisture, providing symptom relief in various situations such as:

* Vaginismus and other sexual dysfunctions related to penetration
* Users of hormonal contraceptives with lubrication loss
* Postpartum and lactational period
* Post antibacterial or antifungal therapies
* During systemic oncological treatments (chemotherapy, radiotherapy, hormone therapy)
* Climacteric (urogenital atrophy)
* Post urogynecological surgeries (correction of urinary incontinence, genital dystopias, etc.)
* Post vulvovaginal abrasive, chemical, laser, or high-frequency therapies
* Post cosmetic and genital rejuvenation therapies

ELIGIBILITY:
Inclusion Criteria:

* Healthy research participants, with an active sexual life;
* Intact skin and mucosa in the test region;
* Participants vaccinated for COVID-19 (Corona virus Disease).
* Agreement to adhere to the study procedures and requirements and attend the institute on the day(s) and time(s) determined for the assessments;
* Ability to consent to participate in the study;
* Menopausal participants of any age, without systemic or topical hormone replacement therapy in the last 6 months
* Presenting mild to moderate vaginal dryness (≥0.5 and <7.5) - according to the Visual Analogic Scale
* Healthy research participants, with an active sex life (at least once a week)

Exclusion Criteria:

* Skin pathology in the area of product application;
* Decompensated Diabetes Mellitus (TBD by the institute together with the sponsor);
* Immune insufficiency;
* Current use of the following topical or systemic medications: corticosteroids, immunosuppressants and antihistamines;
* Skin diseases: vitiligo, psoriasis, atopic dermatitis;
* Previous reaction to the category of the product tested;
* Other illnesses or medications that may directly interfere with the study or put the health of the research participant at risk.
* Have used vaginal moisturizing creams and/or intimate lubricants 5 days before the initial study visit;
* Have had sexual intercourse at least 48 hours before the initial study visit;
* Have been diagnosed with a urogenital or vaginal infection in the last 30 days;
* Have used topical or systemic antibiotics, antifungals, hormone-based creams or treatment for vaginal atrophy in the last 30 days.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Verify the hydration of the cutaneous and genital mucosa after using hyaluronic acid-based vaginal gel | 22 days
  To evaluate the perceived hydration effectiveness, a visual analogue scale will be used, where the minimum value (zero) represents no dryness and the maximum value (ten) represents extremely dryness. Lower scores indicate improved vaginal hydration.
Verify the acceptability of the cutaneous and genital mucosa after using hyaluronic acid-based vaginal gel | 22 days
  To assess skin acceptability, an epithelial integrity questionnaire will be used, where a score, on a 5-point scale, will be assigned after evaluation by the gynecologist. The lowest score will be 1, representing "petechiae before contact" and the maximum score will be 5 with "thin, non-friable mucosa". The higher the score, the healthier and more intact the epithelium will be.

SECONDARY OUTCOMES:
Relief of pruritus after using hyaluronic acid-based vaginal gel | 22 days
  The relief of pruritus assessment will be evaluates through an Visual Analogic Scale. Where the minimum value (zero) represents no pruritus and the maximum value (ten) represents extremely pruritus. Lower scores indicate improvement or absence of vaginal pruritus.
Verify the maintenance of pH after using Hyaluronic Acid when applied under recommended conditions of use through gynecologist follow-up during the use. | 22 days
  pH maintenance will be assessed using reagent strips.
Verify the maintenance of vaginal microbiota after using Hyaluronic Acid when applied under recommended conditions of use through gynecologist follow-up during the use. | 22 days
  Bacterioscopic collection of vaginal contents using a sterile swab. The swabs containing the samples will be placed in test tubes sent to the laboratory for microbiological analysis.

IPD SHARING:
Plan to Share IPD: Undecided